CLINICAL TRIAL: NCT03862469
Title: Premenstrual Hormonal and Affective State Evaluation (PHASE) Project
Acronym: PHASE Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ajna Hamidovic, PharmD, MS, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-1533; R21MH119642 (NIH)
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Premenstrual Dysphoric Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Other)
  Interventions: Procedure: Individualized laboratory test

INTERVENTIONS:
Procedure: Individualized laboratory test — Laboratory test administered between 6 and 2 days prior to the subsequent menstrual cycle.

SUMMARY:
PHASE is designed to evaluate neuroactive hormone trajectories across the menstrual cycle and endocrine, autonomic, and subjective responses to psychosocial stress in women suffering from severe PMS (i.e., premenstrual dysphoric disorder).

DETAILED DESCRIPTION:
Female volunteers will be recruited from the community for participation in this 3-menstrual cycle study. In the first two menstrual cycles, study participants will chart their symptoms and and ovulation. Study participants will continue to perform ovulation testing during their third menstrual cycle in which they will attend one individualized task session and provide 8 serum samples at different timepoints across the menstrual cycle. Primary analyses will contrast neuroactive hormone trajectories across the menstrual cycle and stress reactivity according to study groups (PMDD vs healthy).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-35 years, established by visual inspection of a government-issued ID
* Average menstrual cycle 21-35 days

Exclusion Criteria:

* Lifetime DSM-5 Axis 1 disorder (except anxiety and depression), as documented in the Mental Health Interview
* Current DSM-5 Axis depressive or anxiety disorder, as documented in the Mental Health Interview
* Positive urine drug screen test
* Breath alcohol concentration >0.00%
* Self-reported smoker or carbon monoxide concentration ≥ 6 ppm
* Irregular menstrual cycle
* Current pregnancy (urine test-verified) or lactation, or a plan to become pregnant
* Moderate or high suicide risk
* Shipley IQ (vocabulary standard score) > 80
* Any prescription medications (including hormonal forms of birth control)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajna Hamidovic, PharmD, MS, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Department of Pharmacy Practice, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen AP, Kennedy PJ, Dockray S, Cryan JF, Dinan TG, Clarke G. The Trier Social Stress Test: Principles and practice. Neurobiol Stress. 2016 Nov 12;6:113-126. doi: 10.1016/j.ynstr.2016.11.001. eCollection 2017 Feb. PMID 28229114
- [Background] American College of Obstetricians and Gynecologists. Premenstrual Syndrome. ACOG Practice Bulletin No. 15. Washington, DC: American College of Obstetricians and Gynecologists, 2000.
- [Background] Backstrom T, Sanders D, Leask R, Davidson D, Warner P, Bancroft J. Mood, sexuality, hormones, and the menstrual cycle. II. Hormone levels and their relationship to the premenstrual syndrome. Psychosom Med. 1983 Dec;45(6):503-7. doi: 10.1097/00006842-198312000-00004. PMID 6686333
- [Background] Carlin, J. B., Galati, J. C., & Royston, P. (2008). A new framework for managing and analyzing multiply imputed data in Stata. Stata Journal, 8(1), 49-67.
- [Background] Critchlow DG, Bond AJ, Wingrove J. Mood disorder history and personality assessment in premenstrual dysphoric disorder. J Clin Psychiatry. 2001 Sep;62(9):688-93. doi: 10.4088/jcp.v62n0905. PMID 11681764
- [Background] Cunningham J, Yonkers KA, O'Brien S, Eriksson E. Update on research and treatment of premenstrual dysphoric disorder. Harv Rev Psychiatry. 2009;17(2):120-37. doi: 10.1080/10673220902891836. PMID 19373620
- [Background] Deng D, Pang Y, Duan G, Liu H, Liao H, Liu P, Liu Y, Li S, Chen W, Wen D, Xuan C, Li M. Larger volume and different functional connectivity of the amygdala in women with premenstrual syndrome. Eur Radiol. 2018 May;28(5):1900-1908. doi: 10.1007/s00330-017-5206-0. Epub 2017 Dec 19. PMID 29260367
- [Background] Endicott J, Nee J, Harrison W. Daily Record of Severity of Problems (DRSP): reliability and validity. Arch Womens Ment Health. 2006 Jan;9(1):41-9. doi: 10.1007/s00737-005-0103-y. Epub 2005 Sep 20. PMID 16172836
- [Background] Fischer S, Cleare AJ. Cortisol as a predictor of psychological therapy response in anxiety disorders-Systematic review and meta-analysis. J Anxiety Disord. 2017 Apr;47:60-68. doi: 10.1016/j.janxdis.2017.02.007. Epub 2017 Feb 24. PMID 28273494
- [Background] Hamidovic A, Childs E, Conrad M, King A, de Wit H. Stress-induced changes in mood and cortisol release predict mood effects of amphetamine. Drug Alcohol Depend. 2010 Jun 1;109(1-3):175-80. doi: 10.1016/j.drugalcdep.2009.12.029. Epub 2010 Feb 21. PMID 20176450
- [Background] Howards PP, Schisterman EF, Wactawski-Wende J, Reschke JE, Frazer AA, Hovey KM. Timing clinic visits to phases of the menstrual cycle by using a fertility monitor: the BioCycle Study. Am J Epidemiol. 2009 Jan 1;169(1):105-12. doi: 10.1093/aje/kwn287. Epub 2008 Oct 30. PMID 18974081
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry. 2006 May;63(5):484-9. doi: 10.1001/archpsyc.63.5.484. PMID 16651505
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] Lovick TA. Estrous cycle and stress: influence of progesterone on the female brain. Braz J Med Biol Res. 2012 Apr;45(4):314-20. doi: 10.1590/s0100-879x2012007500044. Epub 2012 Mar 29. PMID 22450372
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Qiao M, Zhang H, Liu H, Luo S, Wang T, Zhang J, Ji L. Prevalence of premenstrual syndrome and premenstrual dysphoric disorder in a population-based sample in China. Eur J Obstet Gynecol Reprod Biol. 2012 May;162(1):83-6. doi: 10.1016/j.ejogrb.2012.01.017. Epub 2012 Feb 28. PMID 22377229
- [Background] Rubinow DR, Schmidt PJ. Gonadal steroid regulation of mood: the lessons of premenstrual syndrome. Front Neuroendocrinol. 2006 Jul;27(2):210-6. doi: 10.1016/j.yfrne.2006.02.003. Epub 2006 May 2. PMID 16650465
- [Background] Schmidt PJ, Nieman LK, Danaceau MA, Adams LF, Rubinow DR. Differential behavioral effects of gonadal steroids in women with and in those without premenstrual syndrome. N Engl J Med. 1998 Jan 22;338(4):209-16. doi: 10.1056/NEJM199801223380401. PMID 9435325
- [Background] Sohda S, Suzuki K, Igari I. Relationship Between the Menstrual Cycle and Timing of Ovulation Revealed by New Protocols: Analysis of Data from a Self-Tracking Health App. J Med Internet Res. 2017 Nov 27;19(11):e391. doi: 10.2196/jmir.7468. PMID 29180346
- [Background] Solis-Ortiz S, Corsi-Cabrera M. Sustained attention is favored by progesterone during early luteal phase and visuo-spatial memory by estrogens during ovulatory phase in young women. Psychoneuroendocrinology. 2008 Aug;33(7):989-98. doi: 10.1016/j.psyneuen.2008.04.003. Epub 2008 Jul 21. PMID 18644678
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Toffol E, Heikinheimo O, Partonen T. Associations between psychological well-being, mental health, and hormone therapy in perimenopausal and postmenopausal women: results of two population-based studies. Menopause. 2013 Jun;20(6):667-76. doi: 10.1097/gme.0b013e318278eec1. PMID 23277355
- [Background] Whooley MA, Grady D, Cauley JA. Postmenopausal estrogen therapy and depressive symptoms in older women. J Gen Intern Med. 2000 Aug;15(8):535-41. doi: 10.1046/j.1525-1497.2000.04029.x. PMID 10940144
- [Background] Yen JY, Wang PW, Su CH, Liu TL, Long CY, Ko CH. Estrogen levels, emotion regulation, and emotional symptoms of women with premenstrual dysphoric disorder: The moderating effect of estrogen receptor 1alpha polymorphism. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Mar 2;82:216-223. doi: 10.1016/j.pnpbp.2017.11.013. Epub 2017 Nov 14. PMID 29146473

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants were retroactively assigned to PMDD versus healthy control cohort after they were diagnosed during their 2nd or 3rd menstrual cycle
Period: Overall Study
Arm/Group | All Participants
Started | 129 (Group assignment is done at the end of the study after all the data is gathered and the participant ends the study. Therefore, it is not known how many participants PER GROUP started the study)
PMDD | 17
Healthy Control | 17
Completed | 34
Not Completed | 95

BASELINE CHARACTERISTICS:
Groups:
- PMDD: PMDD patients
- Controls: Healthy Controls
- Total: Total of all reporting groups
Arm/Group | PMDD | Controls | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, Continuous Population: Age, Continuous
  years | 26.0 (4.8) | 26.36 (5.1) | 26.2 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex: Female, Male Population: Sex: Female, Male
  Participants
    Female | 15 | 14 | 29
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity (NIH/OMB) Population: Ethnicity (NIH/OMB)
  Participants
    Hispanic or Latino | 4 | 4 | 8
    Not Hispanic or Latino | 11 | 9 | 20
    Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race (NIH/OMB) Population: Race (NIH/OMB)
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 5 | 4 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 2 | 4
    White | 5 | 7 | 12
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 1 | 0 | 1
Age of Menarche [Mean (Standard Deviation); unit: years] — Age of Menarche Population: Age of Menarche
  years | 11.4 (1.71) | 12.0 (1.54) | 11.8 (1.60)

OUTCOME MEASURES:

1. Primary Outcome: Hormone Analysis
Description: Cortisol
Time Frame: -20, +20, +30, +40, +50, +65, +90 minutes in the late luteal phase of the menstrual cycle (one day between -1 to -6 days of the subsequent menstrual cycle)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PMDD Patients: PMDD patients
- Healthy Controls: Healthy Controls
Arm/Group | PMDD Patients | Healthy Controls
Number analyzed (Participants) | 15 | 14
ng/mL
  -20 minute timepoint | 70.7 (26.4) | 57.8 (21.9)
  +20 minute timepoint | 114 (53.4) | 97.3 (39.9)
  +30 minute timepoint | 111 (43.6) | 109 (43.6)
  +40 minute timepoint | 97 (48.9) | 100 (32.4)
  +50 minute timepoint | 86.9 (39.4) | 93.3 (29.2)
  +65 minute timepoint | 73.5 (31.6) | 78.4 (24)
  +90 minute timepoint | 70.6 (36.6) | 69 (18.5)

ADVERSE EVENTS:
Time Frame: 12:00 to 15:30 on the day of the session in the late luteal phase of the 2nd menstrual cycle of the study (one day between -1 to -6 days of the subsequent menstrual cycle)
Groups:
- Total: Subjects with and without PMDD
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03862469/Prot_SAP_000.pdf